CLINICAL TRIAL: NCT03618030
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Adult Laboratory Classroom Study to Evaluate the Safety and Efficacy of PRC-063 Compared to Placebo in Adults With ADHD
Brief Title: PRC-063 Adult Laboratory Classroom Study in Adults With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma, Canada (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 063-020
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Results first posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental): PRC-063 25, 35, 45, 55, 70, 85, or 100 mg
  Interventions: Drug: PRC-063 oral capsules
- Placebo Treatment (Placebo Comparator): Matched placebo
  Interventions: Drug: Placebo oral capsules

INTERVENTIONS:
Drug: PRC-063 oral capsules — Daily dose
  Arms: Active Treatment
Drug: Placebo oral capsules — Daily dose
  Arms: Placebo Treatment

SUMMARY:
This is a randomized, double-blind, parallel group, placebo-controlled, dose optimized, phase 3 study to evaluate the safety and efficacy of PRC-063 in the treatment of ADHD in adults

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 18 to 60 years of age
2. Diagnosis of ADHD (any type: combined, predominately hyperactive impulsive type or predominately inattentive type) by a psychiatrist, psychologist, or licensed allied healthcare professional
3. Subject is willing and able to comply with all the protocol requirements.

Exclusion Criteria:

1. Primary and/or comorbid psychiatric diagnosis other than ADHD
2. Has a current or recent history of hypertension, symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems that may place them at increased vulnerability to the sympathomimetic effects of a stimulant drug;
3. Has used any investigational drug within 30 days of the screening visit;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 288 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sailaja Bhaskar, PhD, Study Director — Purdue Pharma, Canada
Locations (8):
- United States (8):
  - Meridien Research Inc., Bradenton, Florida
  - Meridien Research, Lakeland, Florida
  - Meridien Research Inc., Maitland, Florida
  - South Shore Psychiatric Services, Hingham, Massachusetts
  - Center for Psychiatry and Behavioral Medicine, Las Vegas, Nevada
  - Center for Psychiatry and Behavioral Medicine, Durham, North Carolina
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Bayou City Research, Houston, Texas

REFERENCES:
- [Derived] Childress A, Cutler AJ, Marraffino AH, Bhaskar S, Donnelly G. Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Adult Laboratory Classroom Study of the Efficacy and Safety of PRC-063 (Extended-Release Methylphenidate) for the Treatment of ADHD. J Atten Disord. 2022 Apr;26(6):857-869. doi: 10.1177/10870547211025610. Epub 2021 Jun 30. PMID 34189995

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 288 subjects who were screened, 239 subjects were randomized to the double-blind period and were assessed during the full-day adult laboratory classroom (ALC) visit.
Pre-assignment Details: All subjects started on PRC-063 25 mg and were titrated up to his/her optimal dose (25, 35, 45, 55, 70, 85, or 100 mg/day) during the dose optimization period.
  The primary efficacy endpoint compared all doses of PRC-063 combined versus Placebo.
Groups:
- PRC-063 25 mg; PRC-063 35 mg; PRC-063 45 mg; PRC-063 55 mg; PRC-063 70 mg; PRC-063 85 mg; PRC-063 100 mg: PRC-063 oral capsules: Daily dose
Period: Overall Study
Arm/Group | PRC-063 25 mg | PRC-063 35 mg | PRC-063 45 mg | PRC-063 55 mg | PRC-063 70 mg | PRC-063 85 mg | PRC-063 100 mg | Placebo Treatment
Started (Randomized Treatment (in double-blind period) or Last Dose Administered (dose-optimization period)) | 15 | 14 | 21 | 39 | 36 | 27 | 18 | 118
Completed | 3 | 3 | 13 | 30 | 29 | 21 | 14 | 108
Not Completed | 12 | 11 | 8 | 9 | 7 | 6 | 4 | 10

BASELINE CHARACTERISTICS:
Groups:
- Active Treatment: PRC-063 (all doses combined)
  PRC-063 oral capsules: Daily dose
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Placebo Treatment | Total
Number analyzed (Participants) | 121 | 118 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (10.76) | 32.8 (10.95) | 33.6 (10.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 64 | 130
  Male | 55 | 54 | 109
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 21 | 45
  White | 90 | 90 | 180
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Post-dose PERMP-T (Permanent Measure of Productivity - Total Score) Scores Measured During the Full-day Adult Laboratory Classroom Visit
Description: PERMP-T measures the number of completed and number of attempted math problems completed during a 10 minute test. The scale ranges from 0 to 800, with a higher score indicating a better outcome.
Time Frame: Full-day ALC - 13 hours
Population: The full analysis (FA) population was the group of subjects who were randomized and received at least one dose of double-blind study drug, attended the full-day ALC visit evaluation, and had at least one post-dose PERMP-T evaluation during the full-day ALC visit. The primary efficacy endpoint compared all doses of PRC-063 versus Placebo.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Double-Blind Active Treatment: PRC-063 (all doses combined)
  PRC-063 oral capsules: Daily dose
- Double-Blind Placebo Treatment: Matched placebo
  Placebo oral capsules: Daily dose
Arm/Group | Double-Blind Active Treatment | Double-Blind Placebo Treatment
Number analyzed (Participants) | 116 | 113
score on a scale | 302.9 (3.50) | 286.6 (3.52)
Statistical Analysis 1: Comparison: Double-Blind Active Treatment vs Double-Blind Placebo Treatment; The primary efficacy analysis used a mixed-model repeated measures (MMRM) analysis on the full day laboratory classroom PERMP-T scores; Test type: Other; p = .0003, ANOVA

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Safety population: subjects who received at least 1 dose of drug/had at least 1 post-dose safety assessment (N=285 in dose-optimization period; N=239 in double-blind). Since most subjects received multiple dose levels during the dose-optimization period and a subject may have experienced an adverse event which started on one dose level and was ongoing at subsequent dose level(s) during the dose-optimization period, the adverse events for this period are presented for all dose levels combined.
Groups:
- Dose-Optimization: PRC-063 25, 35, 45, 55, 70, 85, or 100 mg oral capsules: Daily dose
- Double-Blind PRC-063 25 mg; Double-Blind PRC-063 35 mg; Double-Blind PRC-063 45 mg; Double-Blind PRC-063 55 mg; Double-Blind PRC-063 70 mg; Double-Blind PRC-063 85 mg; Double-Blind PRC-063 100 mg: PRC-063 oral capsules: Daily dose
Arm/Group | Dose-Optimization | Double-Blind PRC-063 25 mg | Double-Blind PRC-063 35 mg | Double-Blind PRC-063 45 mg | Double-Blind PRC-063 55 mg | Double-Blind PRC-063 70 mg | Double-Blind PRC-063 85 mg | Double-Blind PRC-063 100 mg | Double-Blind Placebo Treatment
All-Cause Mortality (participants affected / at risk) | 0/285 | 0/3 | 0/4 | 0/15 | 0/31 | 0/30 | 0/22 | 0/16 | 0/118
Serious Adverse Events (participants affected / at risk) | 1/285 | 0/3 | 0/4 | 0/15 | 0/31 | 0/30 | 0/22 | 0/16 | 0/118
Other Adverse Events (participants affected / at risk) | 167/285 | 0/3 | 1/4 | 2/15 | 3/31 | 4/30 | 7/22 | 3/16 | 9/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-Optimization (N=285) | Double-Blind PRC-063 25 mg (N=3) | Double-Blind PRC-063 35 mg (N=4) | Double-Blind PRC-063 45 mg (N=15) | Double-Blind PRC-063 55 mg (N=31) | Double-Blind PRC-063 70 mg (N=30) | Double-Blind PRC-063 85 mg (N=22) | Double-Blind PRC-063 100 mg (N=16) | Double-Blind Placebo Treatment (N=118)
Paranoia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-Optimization (N=285) | Double-Blind PRC-063 25 mg (N=3) | Double-Blind PRC-063 35 mg (N=4) | Double-Blind PRC-063 45 mg (N=15) | Double-Blind PRC-063 55 mg (N=31) | Double-Blind PRC-063 70 mg (N=30) | Double-Blind PRC-063 85 mg (N=22) | Double-Blind PRC-063 100 mg (N=16) | Double-Blind Placebo Treatment (N=118)
Headache (Nervous system disorders) | 61 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 61 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 46 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2
Irritability (Psychiatric disorders) | 27 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 26 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Dry Mouth (Gastrointestinal disorders) | 25 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 20 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 17 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 15 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT03618030/Prot_SAP_001.pdf